CLINICAL TRIAL: NCT06824571
Title: Effects of Taurine Supplementation on Repetitive Sprint Performance and Exhaustion Time in College Students Under High-Temperature and High-Humidity Conditions
Acronym: TSPR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xiaodong Cheng (Other)
Responsible Party: Sponsor-Investigator, Xiaodong Cheng, Xian Medical University, Xi'an Medical University
Organization: Xi'an Medical University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: No. 2021A43
Record Dates: First submitted 2025-01-22; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Exercise Performance in Extreme Environments
MeSH Terms: interventions — Taurine

STUDY DESIGN:
Intervention Model Description: This study utilized a single-blind, randomized, crossover-controlled design to evaluate the effects of taurine supplementation at varying doses (6g, 4g, 1g) and placebo on exercise performance under high-temperature and high-humidity conditions. Each participant received all four interventions (high-dose, medium-dose, low-dose, and placebo) in randomized order, with a washout period between treatments to minimize carryover effects. This design allows each participant to serve as their own control, enhancing the precision of the comparisons across conditions.
Who Masked: Participant
Masking Description: The study employed a single-blind design where participants were masked to the intervention assignments. This means that participants were unaware of whether they received high-dose taurine (6g), medium-dose taurine (4g), low-dose taurine (1g), or placebo. The care providers and investigators were aware of the intervention assignments to ensure proper administration and data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High-Dose Taurine Group (6g) (Experimental): Participants in this arm will receive taurine supplementation at a high dose of 6g, dissolved in water, administered 30 minutes prior to exercise.
  High-Dose Taurine Supplementation (6g)
  Interventions: Dietary Supplement: High-Dose Taurine Supplementation (6g)
- Medium-Dose Taurine Group (4g) (Experimental): Participants in this study arm will receive a medium dose of taurine supplementation (4g) in powder form, dissolved in water, administered once 30 minutes prior to exercise. This intervention aims to evaluate the effects of medium-dose taurine on exercise performance, fatigue resistance, and recovery under high-temperature and high-humidity conditions. The study will measure key parameters, including peak power (PP), mean power (MP), fatigue index (FI), exhaustion time (ET), reverse vertical jump values, heart rate (HR), blood lactate (BLA), and ratings of perceived exertion (RPE). This arm is distinguished by the administration of a moderate taurine dosage compared to the high-dose and low-dose groups.
  Interventions: Dietary Supplement: Medium-Dose Taurine Supplementation (4g)
- Low-Dose Taurine Group (1g) (Experimental): Participants in this study arm will receive a low dose of taurine supplementation (1g) in powder form, dissolved in water, administered once 30 minutes prior to exercise. This intervention aims to assess the effects of low-dose taurine on exercise performance, fatigue resistance, and recovery under high-temperature and high-humidity conditions. The study will measure multiple parameters, including peak power (PP), mean power (MP), fatigue index (FI), exhaustion time (ET), reverse vertical jump values, heart rate (HR), blood lactate (BLA), and ratings of perceived exertion (RPE). This arm is distinguished by the administration of a smaller taurine dosage compared to the medium-dose and high-dose groups.
  Interventions: Dietary Supplement: Low-Dose Taurine Supplementation (1g)
- Placebo Group (Placebo Comparator): Participants in this study arm will receive a placebo (inactive substance) in powder form, dissolved in water, administered once 30 minutes prior to exercise. This group serves as the control arm to evaluate the effects of taurine supplementation on exercise performance, fatigue resistance, and recovery under high-temperature and high-humidity conditions. The study will measure key parameters, including peak power (PP), mean power (MP), fatigue index (FI), exhaustion time (ET), reverse vertical jump values, heart rate (HR), blood lactate (BLA), and ratings of perceived exertion (RPE). This arm is distinguished by the administration of an inactive placebo, which contains no taurine, to compare against the taurine intervention arms.
  Interventions: Dietary Supplement: Placebo (0g Taurine)

INTERVENTIONS:
Dietary Supplement: High-Dose Taurine Supplementation (6g) — Participants will receive taurine supplementation at a high dose of 6g. The taurine will be provided in powder form, dissolved in water, and administered 30 minutes prior to exercise. This intervention is designed to evaluate the effects of high-dose taurine supplementation on exercise performance, fatigue resistance, and recovery under high-temperature and high-humidity conditions.
  Arms: High-Dose Taurine Group (6g)
Dietary Supplement: Medium-Dose Taurine Supplementation (4g) — Participants will receive taurine supplementation at a medium dose of 4g. The taurine will be provided in powder form, dissolved in water, and administered 30 minutes prior to exercise. This intervention is designed to evaluate the effects of medium-dose taurine supplementation on exercise performance, fatigue resistance, and recovery under high-temperature and high-humidity conditions.
  Arms: Medium-Dose Taurine Group (4g)
Dietary Supplement: Low-Dose Taurine Supplementation (1g) — Participants will receive taurine supplementation at a low dose of 1g. The taurine will be provided in powder form, dissolved in water, and administered 30 minutes prior to exercise. This intervention is designed to evaluate the effects of low-dose taurine supplementation on exercise performance, fatigue resistance, and recovery under high-temperature and high-humidity conditions.
  Arms: Low-Dose Taurine Group (1g)
Dietary Supplement: Placebo (0g Taurine) — Participants will receive a placebo, consisting of an inactive substance (0g taurine). The placebo will be provided in powder form, dissolved in water, and administered 30 minutes prior to exercise. This intervention serves as a control arm to evaluate the effects of taurine supplementation on exercise performance, fatigue resistance, and recovery under high-temperature and high-humidity conditions.
  Arms: Placebo Group

SUMMARY:
This study is designed to evaluate the effects of acute pre-exercise taurine supplementation at different doses on the performance of college students during exhaustive exercise and subsequent repetitive sprint (RS) activities in a high-temperature, high-humidity environment. Sixteen college students (8 male, 8 female) will participate in a single-blind, randomized, crossover-controlled trial. Participants will be divided into four groups: high-dose taurine (6g), medium-dose taurine (4g), low-dose taurine (1g), and placebo. Key performance metrics such as peak power (PP), mean power (MP), fatigue index (FI), exhaustion time (ET), reverse vertical jump height, heart rate (HR), blood lactate (BLA), and ratings of perceived exertion (RPE) will be measured.

The objective of this study is to assess how taurine supplementation influences exercise performance under these challenging environmental conditions. This study will help to better understand taurine's potential effects on exercise performance and contribute to nutritional strategies for athletes exposed to extreme conditions.

DETAILED DESCRIPTION:
This study is designed to evaluate the effects of taurine supplementation on exercise performance under extreme environmental conditions of high temperature and high humidity. The primary goal is to investigate whether taurine supplementation can enhance performance during exhaustive exercise and subsequent repetitive sprints (RS). Sixteen college students (8 male, 8 female) will participate in a single-blind, randomized, crossover-controlled trial. Participants will be divided into four groups receiving either high-dose (6g), medium-dose (4g), low-dose (1g) taurine supplementation, or placebo.

The study will involve a protocol with exhaustive exercise followed by six repetitive sprints. Performance metrics such as peak power (PP), mean power (MP), and fatigue index (FI) will be recorded. Additionally, physiological parameters, including heart rate (HR) and blood lactate (BLA), as well as subjective measures like ratings of perceived exertion (RPE), will be monitored. A standardized measurement protocol will be used to ensure consistency and accuracy across trials.

ELIGIBILITY:
Inclusion Criteria:

* School students
* Aged between 18 and 28 years
* No exercise-related risk, as indicated by a "no" response to all questions in the Physical Activity Readiness Questionnaire (PAR-Q)
* No taurine-based supplements consumed in the last month.

Exclusion Criteria :

* Individuals who do not meet the inclusion criteria
* Individuals with a history of cardiovascular issues, respiratory problems, or any condition that may impair exercise performance
* Participants who did not provide a "no" response to all questions in the Physical Activity Readiness Questionnaire (PAR-Q)
* Participants who consumed taurine-based supplements in the month preceding the study.

Ages: 20 Days to 26 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Peak Power (Watts) | Measured at the end of each sprint on Day 1 and Day 7.
  Description: Maximum power output during each of the 6 sprints, measured using a cycle ergometer.
  Method of Assessment: Power output will be recorded for each sprint, and the peak value will be identified.
Change from Baseline in Mean Power (Watts) | Measured after all 6 sprints on Day 1 and Day 7.
  Description: Average power output across all 6 sprints, reflecting sustained anaerobic performance.
  Method of Assessment: Power output will be averaged across all sprints.
Change from Baseline in Fatigue Index (%/s) | Measured across all 6 sprints on Day 1 and Day 7.
  Description: Rate of decline in power output across the sprints, representing fatigue resistance.
  Method of Assessment: The decline in power output will be calculated as the difference between the first and last sprint, divided by the time interval.
Change from Baseline in Exhaustion Time (seconds or minutes) | Measured at the point of exhaustion during exhaustive exercise on Day 1 and Day 7.
  Description: The duration participants can sustain exercise before reaching volitional exhaustion.
  Method of Assessment: Time will be recorded from the start of exercise until the participant reaches exhaustion.
Change from Baseline in Blood Lactate Levels (mmol/L) | Measured at baseline (pre-exercise), immediately after exercise, and at specific recovery intervals on Day 1 and Day 7.
  Description: Blood lactate levels will be measured to evaluate metabolic stress and recovery during exercise.
  Method of Assessment: Blood samples will be collected at designated time points during recovery to assess lactate accumulation and clearance.

SECONDARY OUTCOMES:
Change from Baseline in Ratings of Perceived Exertion (RPE) | Measured continuously during exhaustive exercise and repetitive sprint activity on Day 1 and Day 7.
  Description: Participants' perceived physical and mental exertion will be assessed using the Borg Rating of Perceived Exertion Scale.
  Method of Assessment: Participants will rate their exertion on a scale from 6 (no exertion at all) to 20 (maximal exertion).

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong Cheng, PhD, Principal Investigator — Xi'an Medical University
Locations (1):
- Capital University of Physical Education and Sports, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data (IPD) from this study, including anonymized performance metrics, physiological responses, and metabolic data, will be shared with other researchers upon reasonable request. Data will be provided in accordance with applicable ethical and regulatory guidelines to ensure the privacy and confidentiality of study participants. Requests for data access can be made by contacting the principal investigator, Cheng Xiaodong, at chengxiaodong@xiyi.edu.cn.
Supporting Information: SAP
Time Frame: The IPD and supporting information will be made available starting from 6 months after the publication of the study results and will remain available for 5 years.
Access Criteria: The IPD and supporting information will be available to qualified researchers upon request. Access will be granted after a data-sharing agreement is signed to ensure the data will be used responsibly and in accordance with ethical guidelines. Researchers can request access by contacting the Principal Investigator at chengxiaodong@xiyi.edu.cn.

REFERENCES:
- See also: Official website of the Capital University of Physical Education and Sports, where the study was conducted. — https://www.cupes.edu.cn/index.htm

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-09): https://cdn.clinicaltrials.gov/large-docs/71/NCT06824571/Prot_SAP_000.pdf